CLINICAL TRIAL: NCT04854603
Title: The Effect of Dairy Products With Reduced Added Sugar Content on Blood Glucose, Satiety and Food Intake
Brief Title: Dairy Products With Reduced Sugar and Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Saint Vincent University (Other)
Responsible Party: Principal Investigator, Bohdan Luhovyy, Associate Professor, Mount Saint Vincent University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2019-202-01
Record Dates: First submitted 2021-04-10; First posted 2021-04-22 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Blood Glucose, High; Metabolic Disease; Overweight and Obesity
Keywords: Sugar intake; Sweeteners; Diabetes; Obesity; Sweetened food products; Chocolate milk
MeSH Terms: conditions — Metabolic Diseases; Overweight; Obesity; Diabetes Mellitus | interventions — Food

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Treatments will be blinded. The Investigator will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Chocolate milk with a regular added sugar content (Experimental): Dairy product with a regular sugar content
  Interventions: Other: Food
- Chocolate milk with a reduced added sugar content (Experimental): Dairy product with a reduced sugar content
  Interventions: Other: Food
- Yogurt with a regular added sugar content (Experimental): Dairy product with a regular sugar content
  Interventions: Other: Food
- Yogurt with a reduced added sugar content (Experimental): Dairy product with a reduced sugar content
  Interventions: Other: Food
- Energy-free control (Experimental): Potable water
  Interventions: Other: Food

INTERVENTIONS:
Other: Food — Dairy products with regular and reduced sugar content and water control.

SUMMARY:
Dairy products represent an important food group in human nutrition as a source of calcium, protein, functional fats and low-glycaemic sugar lactose. While traditionally consumed natural milk and yogurt have low sugar content, many flavoured liquid dairy products such as chocolate milk, or fermented products such as yogurt have added sugar. Our recent studies have shown that the partial reduction of added sugar in chocolate milk and yogurt is not associated with any inferior sensory characteristics such as taste and pleasantness compared to their full-sugar counterparts. The current project will investigate whether the liquid dairy products with reduced sugar content (value-added products) have any benefits on blood glucose control in humans.

ELIGIBILITY:
Inclusion Criteria:

* 19-35 y males and females, non-smokers

Exclusion Criteria:

* having any diseases, irregular menses in females, smoking (all types), taking medications known to influence blood glucose control, skipping breakfast, and having emotional, or learning problems that would affect their ability to participate in the study as required. Individuals with known food allergies and lactose intolerance will be also excluded.

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Blood glucose | 0-120 minutes
  The concentration of blood glucose
Insulin | 0-120 minutes
  The concentration of blood glucose

SECONDARY OUTCOMES:
Satiety | 0-120 minutes
  The components of average subjective appetite including desire to eat, hunger, fullness, and a prospective food consumption measured with 100mm visual analogue scales.
Food intake | 120 minutes
  Energy intake with an ad libitum meat at 120 minutes
Thirst | 0-120 minutes
  The subjective perception of thirst measured with 100mm visual analogue scales containing the question "How thirsty do you feel?" and two statements on each pole of 100mm line: "Not thirsty at all" (0mm) and "As thirsty as I have ever felt" (100mm).
Physical comfort | 0-120 minutes
  The subjective feeling of wellness and gastrointestinal discomfort parameters including the feeling of nausea, stomach cramps, flatulency, diarrhea and a subjective feeling of wellness, each measured with 100mm visual analogue scales.
Food pleasantness | at 0 and 120 minutes
  The perception of pleasantness of the treatments (0 min) and a test meal (at 120 min) will be measured with 100mm visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Bohdan Luhovyy, PhD, Principal Investigator — Mount Saint Vincent University
Locations (1):
- Mount Saint Vincent University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No